CLINICAL TRIAL: NCT02063776
Title: The Effects of Haemodiafiltration (HDF) vs Conventional Haemodialysis (HD) on Growth and Cardiovascular Markers in Children - 3H (HDF, Hearts and Height) Study
Brief Title: Haemodiafiltration vs Conventional Haemodialysis in Children
Acronym: 3H
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13NU02
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Children; Haemodialysis; Haemodiafiltration
Keywords: Haemodiafiltration (HDF); Haemodialysis (HD); Children; Carotid intima media thickness; Pulse wave velocity; Height standard deviation score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children on HDF
- Children on conventional HD

SUMMARY:
Children on conventional haemodialysis (HD) die of heart disease. Also, they can be malnourished and short. Haemodiafiltration (HDF) is a newer type of dialysis that achieves better removal of toxins and excess fluid than HD. On HDF, adults have a longer survival and children show improved growth, but mechanisms are not understood.

We will follow children in the UK and Europe to compare HDF and HD. We will monitor growth, heart and blood vessel scans, blood markers and quality of life. If the 3H (HDF-Hearts-Height) study shows reduced cardiovascular morbidity and better growth, HDF may be adopted as the preferred type of dialysis in children.

DETAILED DESCRIPTION:
Background: Children on conventional haemodialysis (HD) have a 1000-fold higher mortality than their healthy peers and can have malnutrition and growth retardation. Haemodiafiltration (HDF) achieves better clearance of uraemic solutes across a wide molecular-weight range and performs greater ultrafiltration than conventional HD. Randomised controlled trials in adults have shown 35-45% improved survival and reduced cardiovascular mortality on HDF with high convection volumes. Excellent catch-up growth has been demonstrated in children on HDF, but mechanisms are poorly understood.

Hypothesis: HDF improves the cardiovascular risk profile, growth and quality of life (QoL) compared to conventional HD. Primary outcome measures are carotid intima-media thickness (cIMT) and height standard deviation score (SDS).

Plan of investigation: Incident and prevalent patients on HDF or HD who are expected to remain on dialysis for >6-months and who have a single pool Kt/v>1.2 will be compared in a 1:1 study design. Anthropometric measures (height SDS, body mass index SDS) and QoL questionnaires will be monitored at baseline and 6-monthly. Cardiovascular measures (cIMT, pulse wave velocity, left ventricular mass index and 24-hour BP) will be measured annually. 6-monthly blood tests will measure nutritional biomarkers, mineral dysregulation, inflammation and middle-molecule clearance. Outcome measures will be standardised to the convective clearance dose per m2 body surface area. Recruitment will continue for 2½ years with minimum follow-up of 6-months.

Children will be recruited from all UK dialysis units, but small patient numbers (10-12/year) necessitate collaborations with European centres. HDF and HD patients across Europe who are part of the Cardiovascular Comorbidity in Childhood CKD (4C) study will be included and vascular scans will be captured from this study. From ESPN/ERA-EDTA registry data we estimate ~100 children on HDF over the study period.

Outcomes: If the 3H (HDF-Hearts-Height) study shows that HDF reduces cardiovascular morbidity and improves growth it may lead to HDF being adopted as the standard for in-centre dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. All children 5 - 21 years age undergoing HDF in paediatric dialysis centres (incident and prevalent patients)
2. Age-matched HD patients
3. Prevalent HDF and HD patients must achieve a single pool Kt/v>1.2 in the month preceding recruitment

Exclusion Criteria:

1. Children in whom a living donor kidney transplant is planned within 6-months of start of dialysis

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * HDF patients will be compared with age-matched HD patients in a 1:1 study design.
  * Children will be recruited from paediatric dialysis units within the UK and also centres in Europe, through the 4C-study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2017-05 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
1. Change in carotid artery intima-media thickness (cIMT) standard deviation score (SDS) | 12 months
Change in height SDS | 12 months

SECONDARY OUTCOMES:
For nutritional status 1. Body mass index SDS 2. Markers of appetite regulation and nutritional status | 6 months
For cardiovascular status 1. 24-hour mean arterial BP SDS 2. Left ventricular mass index 3. Pulse wave velocity SDS 4. Biomarkers of cardiovascular disease | 12 months
Quality of life (QoL) questionnaires | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rukshana C Shroff, MD FRCPCH PhD, Study Chair — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Rukshana Shroff, London, United Kingdom

REFERENCES:
- [Derived] Shroff R, Bayazit A, Stefanidis CJ, Askiti V, Azukaitis K, Canpolat N, Agbas A, Anarat A, Aoun B, Bakkaloglu S, Bhowruth D, Borzych-Duzalka D, Bulut IK, Buscher R, Dempster C, Duzova A, Habbig S, Hayes W, Hegde S, Krid S, Licht C, Litwin M, Mayes M, Mir S, Nemec R, Obrycki L, Paglialonga F, Picca S, Ranchin B, Samaille C, Shenoy M, Sinha M, Smith C, Spasojevic B, Vidal E, Vondrak K, Yilmaz A, Zaloszyc A, Fischbach M, Schaefer F, Schmitt CP. Effect of haemodiafiltration vs conventional haemodialysis on growth and cardiovascular outcomes in children - the HDF, heart and height (3H) study. BMC Nephrol. 2018 Aug 10;19(1):199. doi: 10.1186/s12882-018-0998-y. PMID 30097064
- [Derived] Agbas A, Canpolat N, Caliskan S, Yilmaz A, Ekmekci H, Mayes M, Aitkenhead H, Schaefer F, Sever L, Shroff R. Hemodiafiltration is associated with reduced inflammation, oxidative stress and improved endothelial risk profile compared to high-flux hemodialysis in children. PLoS One. 2018 Jun 18;13(6):e0198320. doi: 10.1371/journal.pone.0198320. eCollection 2018. PMID 29912924